CLINICAL TRIAL: NCT01391767
Title: Histologic Evaluation of Healing Following Tooth Extraction With Ridge Preservation Using NuOss XC and NuOss Particulate
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Collaborators: ACE Surgical Supply, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Nuoss-15852
Record Dates: First submitted 2011-07-01; First posted 2011-07-12 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Oral Ridge Preservation
Keywords: Ridge Preservation; Dental Implant; Histology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Hard tissue histological evaluation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NuOss XC: Bone grafting material used in this group will be NuOss XC.
  Interventions: Device: NuOss XC
- NuOss Particulate: Bone grafting material used in this group will be NuOss Particulate.

INTERVENTIONS:
Device: NuOss XC — NuOss XC is a bone grafting material that will be placed in extraction socket site.
  Groups: NuOss XC

SUMMARY:
This study histologically evaluates sites grafted with NuOss XC using ridge preservation techniques prior to placement of dental implants. Sites grafted with NuOss XC (bovine bone mineral with self-expanding collagen) will be compared to sites grafted with NuOss particulate (bovine bone mineral).

DETAILED DESCRIPTION:
Patients presenting to the University of Oklahoma College of Dentistry Graduate Periodontics Clinic who are treatment planned for tooth extraction and placement of dental implant(s) will be interviewed for possible participation in the study. Forty extraction sites will be included in this study to provide statistical significance.

The ridge preservation sites, using either NuOss XC or NuOss particulate, will be selected randomly. The first site will be selected using the flip of a coin. Thereafter, every other site will be grafted using NuOs XC. The ridge preservation procedure will involve tooth extraction with as little trauma as possible to preserve all four bony socket walls, curettage of the socket to remove all periodontal ligament fibers and granulation tissue, placement of the graft material into the socket and coverings the graft material with long-lasting collagen membrane. Facial and lingual mucoperiosteal flaps will be elevated to facilitate securing of the membrane with long-lasting absorbable sutures. Patient will be given prescriptions for analgesics and antibiotics as necessary.

ELIGIBILITY:
INCLUSION CRITERIA:

* may be either male or female
* must be between 18 and 64 years old
* must be of sufficiently good health to undergo routine dental treatment, including the surgical procedures associated with tooth extraction and placement of NuOss XC or NuOss particulate
* must agree to remain in study for 6 months after ridge preservation (grafting)
* must be able to physically, emotionally, and financially undergo the surgical and restorative (implant replacement) procedures planned.
* must not have medical conditions that preclude the removal of indicated teeth and placement of NuOss XC or NuOss particulate
* must have at least one single-rooted tooth to be extracted
* must consent to tooth extractions, socket augmentation and implant placement
* Patients with or without dental insurance

Exclusion Criteria:

* have any requirements for antibiotic premedication for heart murmurs, artificial joints, or any other condition
* have a history of significant heart, stomach, liver, kidney, blood, immune system or other organ impairment or systemic disease that would prevent their undergoing the proposed treatment
* smoke ≥ 10 cigarettes per day or use other tobacco products
* have a religious or philosophical aversion to having processed bovine bone or collagen used in their mouth
* have taken any investigational drugs anytime in the previous month
* have dental conditions likely to require treatment, necessitating exit from the study such as deep caries, abscesses, or moderate-severe periodontal disease(s).
* have sockets that do not have four bony walls intact.
* cannot comply with treatment and follow-up visits for 6 months
* have had significant radiation exposure (occupational, therapeutic, diagnostic).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Periodontal Clinic Population at the University of Oklahoma College of Dentistry
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Histological analysis: All sections removed from the osteotomy (hole where implant will be placed) at time of implant placement to be evaluated by a single evaluator, using a semi-quantitative scoring system | 12-18 months
  Histological processing: Specimens to be trimmed and embedded in methyl methacrylate (MMA). One hematoxylin and eosin (H&E) stained section, and one Goldner's trichrome-stained section to be taken from each block in a longitudinal plane through the approximate center of each defect.
  Goldner's trichrome-stained slides to be scored for the presence of bone and bone marrow as a percent of the total defect area.
  H&E-stained slides to be used to evaluate residual collagen and residual bone mineral as a percent of the total defect area.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Carson, DMD, MS, Principal Investigator — University of Oklahoma College of Dentistry
Locations (1):
- University of Oklahoma College of Dentistry, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Jemt T, Lekholm U. Implant treatment in edentulous maxillae: a 5-year follow-up report on patients with different degrees of jaw resorption. Int J Oral Maxillofac Implants. 1995 May-Jun;10(3):303-11. PMID 7615326
- [Background] Iasella JM, Greenwell H, Miller RL, Hill M, Drisko C, Bohra AA, Scheetz JP. Ridge preservation with freeze-dried bone allograft and a collagen membrane compared to extraction alone for implant site development: a clinical and histologic study in humans. J Periodontol. 2003 Jul;74(7):990-9. doi: 10.1902/jop.2003.74.7.990. PMID 12931761